CLINICAL TRIAL: NCT05121272
Title: Fatigue and Cognitive Demand With Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 13406
Record Dates: First submitted 2021-09-03; First posted 2021-11-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fatigue
Keywords: sex difference; aging
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- young men (Experimental): Individuals will participate in 1 familiarization and 3 test sessions
  Interventions: Behavioral: cognitive task
- young women (Experimental): Individuals will participate in 1 familiarization and 3 test sessions
  Interventions: Behavioral: cognitive task
- older men (Experimental): Individuals will participate in 1 familiarization and 3 test sessions
  Interventions: Behavioral: cognitive task
- older women (Experimental): Individuals will participate in 1 familiarization and 3 test sessions
  Interventions: Behavioral: cognitive task

INTERVENTIONS:
Behavioral: cognitive task — cognitive task

SUMMARY:
This study will determine the influence of a cognitive task performed during fatiguing contractions.

DETAILED DESCRIPTION:
Individuals will participate in one familiarization session followed by 3 randomized experimental sessions (crossover design).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged between 18-35 and 65-90

Exclusion Criteria:

* Metal implants or joint replacement. neuromuscular disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
force | Each session will take approximately 2-3 hours (total of 4 test sessions)
  Change in force of the arm muscles will be evaluated with a custom made device during each test session
anxiety levels | Each session will take approximately 2-3 hours (total of 4 test sessions
  changes in anxiety levels quantified with a questionnaire
arterial pressure | Each session will take approximately 2-3 hours (total of 4 test sessions
  changes in arterial pressure will be quantified with a non-invasive device (finometer)
fatigue | Each session will take approximately 2-3 hours (total of 4 test sessions
  changes in fatigue will be assessed with questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Pereira, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma, Norman, Oklahoma, United States